CLINICAL TRIAL: NCT06078852
Title: Longitudinal Interventional Study on Diaphragmatic Ultrasound in Facioscapulohumeral Dystrophy (FSHD) Patients
Brief Title: Longitudinal Study on Diaframmatic Ultrasound in FSHD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5778
Record Dates: First submitted 2023-07-10; First posted 2023-10-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-11

CONDITIONS: FSHD1; FSHD2
MeSH Terms: interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FSHD patients (Experimental): Patients with genetically confirmed FSHD undergoing routine neurological and pneumological follow-up, who will be assessed with diaphragmatic ultrasound and standard pulmonary function tests at baseline and at 12 months.
  Interventions: Other: Diaphragmatic ultrasound; Other: Pulmonary function test

INTERVENTIONS:
Other: Diaphragmatic ultrasound — Ultrasound evaluation of diaphragm thickness, contractility, and excursion in semi-supine and sitting positions.
Other: Pulmonary function test — Routine spirometry, body plethysmography (FRC, TLC), maximal inspiratory/expiratory pressures (MIP, MEP), and nocturnal oximetry.

SUMMARY:
The goal of this prospective, longitudinal, single-center study is to describe respiratory function in patients affected by FSHD at baseline and after one year using both diaphragmatic ultrasound and pulmonary function test. The primary questions this study aims to answer are:

1. How does respiratory function assessed by diaphragmatic ultrasound and pulmonary function tests change over 12 months in FSHD patients?
2. How accurate is diaphragmatic ultrasound in detecting respiratory abnormalities in these patients compared to pulmonary function tests?
3. What is the relationship between ultrasound and functional indices, and how do these indices correlate with demographic, clinical, and genetic data?

To achieve this, we will enroll a cohort of 34 patients affected by FSHD, and each of them will undergo a comprehensive neurological examination, body plethysmography, measurement of maximal inspiratory pressure (MIP) and maximal espiratory pressure (MEP) and nocturnal oximetry at baseline and after 12 months.

DETAILED DESCRIPTION:
Respiratory involvement is a recognized but underexplored manifestation of facioscapulohumeral muscular dystrophy (FSHD), reported in up to half of affected individuals. It is primarily related to weakness of the diaphragm and abdominal muscles, as well as to possible thoracic deformities. Traditional spirometric tests may underestimate early or mild inspiratory abnormalities, limiting their sensitivity for clinical monitoring. Diaphragmatic ultrasound has recently emerged as a promising tool to assess both trophism and contractility of the diaphragm. To date, only one small cross-sectional study has applied this technique in FSHD, showing reduced diaphragmatic parameters compared to controls, and no longitudinal data are currently available.

This study aims to provide the first prospective evaluation of diaphragmatic ultrasound in a cohort of genetically confirmed FSHD patients, with assessments performed at baseline and after one year of follow-up. By combining diaphragmatic ultrasound with standardized pulmonary function tests, body plethysmography, and respiratory muscle strength measurements, the study will comprehensively characterize respiratory involvement in FSHD and evaluate the potential role of ultrasound-derived indices as sensitive biomarkers.

The study design allows for the correlation of ultrasound findings with clinical and demographic characteristics, including disease duration, genetic features, and severity scores, as well as with conventional pulmonary outcomes. The longitudinal approach will clarify the ability of ultrasound to detect early or progressive respiratory impairment and its potential to complement or surpass routine respiratory function tests.

Ultimately, this project seeks to establish diaphragmatic ultrasound as a feasible and reproducible tool for the monitoring of respiratory function in FSHD. The expected results may inform the development of improved clinical guidelines for respiratory surveillance and contribute to early identification of patients who may benefit from targeted interventions, such as respiratory physiotherapy or non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FSHD, genetically confirmed.
* Adult patients (18 years or older)
* Signature from the patient on the written informed consent document

Exclusion Criteria:

- Medical history of neck and mediastinal trauma and/or surgery and/or radiation therapy (e.g. total thyroidectomy, mastectomy) with evidence of phrenic nerve injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
One-year evaluation of the ultrasound diaphragmatic trophism | At enrollement and one year -follow-up
  Diaphragmatic thickness (DT) after a normal expiration (basal-DT) and after a maximal inspiration (max-DT)
One-year evaluation of the ultrasound diaphragmatic contractility | At enrollement and one year -follow-up
  Diaphragmatic thickening after a maximal inspiration determined as the difference between max-DT and basal-DT
One-year evaluation of the ultrasound diaphragmatic contractility (as ratio) | At enrollement and one year -follow-up
  Diaphragmatic thickening after a maximal inspiration determined as the ratio of difference between max-DT and basal-DT to basal-DT
One-year evaluation of the ultrasound diaphragmatic excursion | At enrollement and one year -follow-up
  Diaphragmatic excursion after a maximal inspiration

CONTACTS AND LOCATIONS:
Overall Officials: Ricci Enzo, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy